CLINICAL TRIAL: NCT01394770
Title: Cardiovascular Events in Hypertensive Hemodialysed Patients: Aliskiren Versus Amlodipine. A Randomized, Double-blind Study.
Brief Title: Aliskiren or Amlodipine in Hypertensive Hemodialysed Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Gennaro Cice, MD, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AL-AM dial
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Hypertension; Dialysis
Keywords: hypertension; dialysis; aliskiren; amlodipine; outcome
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Experimental)
  Interventions: Drug: Aliskiren
- Amlodipine (Active Comparator)
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 mg for 1 month with forced uptitration to 300 mg compared in parallel group with amlodipine 5 mg with forced uptitration to 10 mg
  Other Names: Rasilez, Norvasc

SUMMARY:
Hypertensive haemodialysis patients are at high risk for cardiovascular events. This study was undertaken to ascertain whether aliskiren, a direct renin inhibitor, compared with amlodipine, a calcium channel blocker, reduces mortality and cardiovascular events in these high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysed patients
* predialytic blood pressure greater or equal to 140/90 mmHg

Exclusion Criteria:

* history of heart failure
* history of ischemic heart disease
* severe aortic stenosis
* known allergy to aliskiren or amlodipine
* severe disorders of liver function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
composite end-point of: all-cause mortality; cardiac event including myocardial infarction, need for coronary angioplasty or coronary bypass surgery, ischaemic stroke | 30 months

SECONDARY OUTCOMES:
composite end-point of: all-cause hospitalization, new-onset heart failure,new-onset atrial fibrillation | 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Second Univesity of Naples, Naples, Italy

REFERENCES:
- [Derived] Mugendi GA, Mutua FM, Natale P, Esterhuizen TM, Strippoli GF. Calcium channel blockers for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 Oct 1;10(10):CD011064. doi: 10.1002/14651858.CD011064.pub2. PMID 33000470